CLINICAL TRIAL: NCT00669019
Title: A Phase 2 Study of AZD0530 in Metastatic Melanoma
Brief Title: Saracatinib in Treating Patients With Stage III or Stage IV Melanoma That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00193; N01CM62201 (NIH); CDR0000594729 (Registry Identifier: PDQ (Physician Data Query)); 16077A
Record Dates: First submitted 2008-04-26; First posted 2008-04-29 (Estimated); Results first posted 2014-01-27 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-01

CONDITIONS: Recurrent Melanoma; Stage IIA Melanoma; Stage IIB Melanoma; Stage IIC Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — saracatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Saracatinib (Experimental): Patients receive saracatinib 175 mg oral once daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: saracatinib

INTERVENTIONS:
Drug: saracatinib
  Other Names: AZD0530

SUMMARY:
This phase II trial is studying how well saracatinib works in treating patients with stage III or stage IV melanoma that cannot be removed by surgery. Saracatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the Src kinase inhibitor, AZD0530 (saracatinib), has single agent clinical activity in patients with advanced melanoma.

II. To determine whether this drug will increase progression-free survival of these patients from 3 months to 4.5 months.

SECONDARY OBJECTIVES:

I. To determine whether this drug may inhibit the activation of peripheral blood T cells analyzed ex vivo.

OUTLINE:

Patients receive saracatinib orally (PO) once daily (QD) in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic melanoma

  * Stage IV or unresectable stage III disease
* Measurable disease, defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded) as ≥ 20 mm by conventional techniques or as ≥ 10 mm by spiral computed tomography (CT) scan
* No known brain metastases
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 12 weeks
* White blood cell (WBC) ≥ 3,000/mcL
* Absolute neutrophil count (ANC) ≥ 1,500/mcL
* Platelet count ≥ 100,000/mcL
* Hemoglobin ≥ 9 g/dL
* Total bilirubin normal
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Proteinuria ≤ 1+ by dipstick OR 24-hour urine protein ≤ 1 g
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception prior to study until completion of study treatment
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD0530
* No QTc prolongation (defined as a QTc interval ≥ 480 msecs) or other significant electrocardiogram (ECG) abnormalities
* No poorly controlled hypertension (e.g., systolic blood pressure [BP] of ≥ 140 mm Hg or diastolic BP of ≥ 90 mm Hg)
* No condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation), prior surgical procedures affecting absorption, or active peptic ulcer disease that impairs the ability to swallow AZD0530 tablets
* No intercurrent cardiac dysfunction including, but not limited to, any of the following:

  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
* No recent history of ischemic heart disease including myocardial infarction
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
* No other malignancy within the past 5 years, except definitively treated, localized, nonmelanoma skin cancer or low-grade cervical neoplasm
* At least 4 weeks since prior and no more than one prior treatment regimen for advanced disease
* No prior kinase inhibitor with activity against Src kinases for metastatic melanoma
* More than 4 weeks since prior luteinizing hormone-releasing hormone agonists
* No concurrent combination antiretroviral therapy for human immunodeficiency virus (HIV)-positive patients
* No concurrent prohibited cytochrome P450 3A4 (CYP3A4)-active agents or substances

  * Prohibited drugs should be discontinued 7 days prior to the administration of the first dose of AZD0530 and for 7 days following discontinuation of AZD0530
* No other concurrent investigational agents or commercial therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gajewski, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at five sites in the United States between August 2008 and September 2009.
Groups:
- Saracatinib: Patients receive saracatinib 175 mg oral, once daily in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Saracatinib
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Saracatinib
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 63 [25 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 23
Performance Status [Number; unit: participants] — ECOG performance status scores on a scale of 0-5, higher is worse
  0 = Fully active, able to carry on all pre-disease performance without restriction
  1. = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about > 50% of waking hours
  3. = Capable of only limited self-care, confined to bed/chair more than 50% of waking hours
  4. = Completely disabled. Cannot carry on any self-care. Totally confined to bed/chair
  5. = Dead
  participants
    0 | 13
    1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Response will be evaluated in this study using the Response Evaluation Criteria in Solid Tumors (RECIST). A sum of the longest diameter (LD) for all target lesions will be calculated and reported as the baseline sum LD. The baseline sum LD will be used as reference by which to characterize the objective tumor response. Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum LD; Objective response = CR + PR.
  CT scans will be performed at baseline and every 4-8 weeks while on study.
Time Frame: Up to 25 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Saracatinib
Number analyzed (Participants) | 23
percentage of participants | 0 [0 to 14.8]

2. Secondary Outcome: Progression-free Survival
Description: Progression will be evaluated in this study using the RECIST criteria (the appearance of new lesions and/or at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study). Progression-free survival time was calculated as the time from treatment start to date of progression or death, whichever comes first.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Saracatinib
Number analyzed (Participants) | 23
weeks | 7.4 [7.0 to 7.9]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored over the course of treatment
Description: treatment related adverse events are reported
Arm/Group | Saracatinib
Serious Adverse Events (participants affected / at risk) | 1/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saracatinib (N=23)
Creatinine increased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saracatinib (N=23)
Fatigue (General disorders) | 19
Hyperglycemia (Metabolism and nutrition disorders) | 17
Anemia (Blood and lymphatic system disorders) | 15
Diarrhea (Gastrointestinal disorders) | 13
Anorexia (Metabolism and nutrition disorders) | 11
Hypocalcemia (Metabolism and nutrition disorders) | 10
Nausea (Gastrointestinal disorders) | 11
Hyponatremia (Metabolism and nutrition disorders) | 9
Aspartate aminotransferase increased (Investigations) | 7 — Aspartate aminotransferase/alanine aminotransferase increased
Vomiting (Gastrointestinal disorders) | 5
Platelet count decreased (Investigations) | 5 — Thrombocytopenia
Lymphocyte count decreased (Investigations) | 7 — Lymphopenia

LIMITATIONS AND CAVEATS:
Trial was designed with a maximum target accrual of 37 patients. Per protocol, the trial was stopped after the first stage based on an interim analysis of the response rate among the first 23 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less